CLINICAL TRIAL: NCT07036172
Title: A Multicenter, Randomized, Open-label, Parallel-controlled Phase III Clinical Study Comparing the Efficacy and Safety of Semaglutide Injection and WEGOVY® in Chinese Obese Patients
Brief Title: Efficacy and Safety of Semaglutide Injection Vs WEGOVY® in Chinese Obese Patients
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hangzhou Zhongmei Huadong Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HDM1702-301
Record Dates: First submitted 2025-06-16; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Obesity Control
MeSH Terms: interventions — semaglutide

STUDY DESIGN:
Masking Description: Statistician, data manager and medical monitor are masked to the randomized allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HDM1702 (Experimental)
  Interventions: Drug: HDM1702
- WEGOVY® (Active Comparator)
  Interventions: Drug: Wegovy ®

INTERVENTIONS:
Drug: HDM1702 — Initiate at a once weekly dose of 0.25 mg and followed a fixed-dose escalation regimen, with dose increases every 4 weeks (to doses of 0.5, 1.0, 1.7 and 2.4 mg per week) aiming at reaching the maintenance dose of 2.4 mg at week 16.
  Arms: HDM1702
Drug: Wegovy ® — Initiate at a once weekly dose of 0.25 mg and followed a fixed-dose escalation regimen, with dose increases every 4 weeks (to doses of 0.5, 1.0, 1.7 and 2.4 mg per week) aiming at reaching the maintenance dose of 2.4 mg at week 16.
  Arms: WEGOVY®

SUMMARY:
This is a 48-week randomized, open-label, parallel-controlled biosimilar comparison study comparing the efficacy, safety and immunogenicity of the investigational drug and WEGOVY® in patients with obesity. Eligible participants will be screened and randomized to the experimental group and the active comparator group at a ratio of 1:1 , semaglutide injection or WEGOVY® injection will be given once weekly for 44 weeks, following by a safety follow up of 4 weeks. All participants received a lifestyle intervention that involved counselling on diet and physical activity.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged ≥18 years and ≤75 years at the time of signing informed consent；
2. BMI ≥28 kg/m2；
3. A self-reported change in body weight no more than 5% within 90 days before screening.

Exclusion Criteria:

1. History of type 1 and type 2 diabetes;
2. Previous or planned (during the trial period) obesity treatment with surgery or a weight-loss device;
3. History or presence of chronic or acute pancreatitis;
4. Personal or first-degree relative(s) history of multiple endocrine neoplasia type 2 or medullary thyroid carcinoma;
5. A history or presence of suspected depression or other mental disorders;
6. Patient Health Questionnaire-9 score of ≥15 at screening
7. Uncontrolled hypertension, any of the following: myocardial infarction, stroke, hospitalisation for unstable angina, or transient ischaemic attack within the past 6 months prior to screening;
8. History of malignant neoplasms within the past 5 years prior to screening;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male or female aged 18 years to 75 years (inclusive) at the time of signing the informed consent
Enrollment: 460 (Estimated)
Dates: Start 2025-01-03 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
The percentage change in body weight from baseline to week 44 | week 44

SECONDARY OUTCOMES:
The proportion of participants reaching a body weight loss of at least 5%, 10% and 15% at week 44 | week 44
Change in waist circumference, body weight and BMI at week 44 | week 44
Change in blood pressure and lipids at week 44 | week 44
Adverse events | week 44
ADA and NAb | week 44

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, China